CLINICAL TRIAL: NCT05197322
Title: NEOPRISM-CRC : Neoadjuvant Pembrolizumab Stratified to Tumour Mutation Burden for High Risk Stage 2 or Stage 3 MMR-deficient Colorectal Cancer
Brief Title: NEOadjuvant PembRolizumab In Stratified Medicine - ColoRectal Cancer
Acronym: NEOPRISM-CRC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Sharp (Industry); Foundation Medicine (Industry); University College London (UCL) Cancer Institute (Other); University of Leeds (Other); University College London Hospitals (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCL/127464
Record Dates: First submitted 2021-12-14; First posted 2022-01-19 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: Adenocarcinoma of the Colon
MeSH Terms: conditions — Colonic Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: Open label, 2 arm phase II trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tumour Mutation Burden high or medium (or MSI-High) (Other): Patients will one cycle of pembrolizumab 200 mg IV (a cycle is 21 days). Prior to cycle 2 the result of the FOUNDATIONONE®CDx test or FOUNDATIONONE® Liquid CDx should be available and patients will continue their treatment as follows:
  TMB-high (defined as ≥20 mutations per Mb) or medium (defined as 6-19 mutations per Mb); FOUNDATIONONE®CDx or FOUNDATIONONE® Liquid CDx test (or MSI-H if FOUNDATIONONE®CDx or FOUNDATIONONE® Liquid CDx test is not evaluable):
  * A further two cycles of pembrolizumab 200 mg IV every 21 days
  * Planned surgery to remove the CRC 4 - 6 weeks after last dose of pembrolizumab
  Interventions: Drug: Pembrolizumab
- Tumour Mutation Burden low or unevaluable (Other): Patients will one cycle of pembrolizumab 200 mg IV (a cycle is 21 days). Prior to cycle 2 the result of the FOUNDATIONONE®CDx or FOUNDATIONONE® Liquid CDx test should be available and patients will continue their treatment as follows:
  TMB-low (defined as ≤5 mutations per Mb); FOUNDATIONONE®CDx or FOUNDATIONONE® Liquid CDx OR if FOUNDATIONONE test and MSI result by PCR are both not evaluable):
  • Planned surgery to remove the CRC 4 - 6 weeks after last dose of pembrolizumab
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — Dose: 200mg by IV infusion on Day 1 of each treatment cycle

SUMMARY:
Colorectal cancer (CRC) is the 2nd to 3rd most common malignant disease in developed countries, with over 1 million new cases and 500,000 deaths worldwide each year. The primary treatment for early stage CRC is surgery to remove the tumour, which is possible in 80% of patients. Even after surgery up to half of patients will develop recurrence or spread of the disease (metastases) which is incurable. Survival after 5 years is approximately 14% for patients with metastatic disease. Clinical trials using immunotherapy drugs called 'immune checkpoint inhibitors' have shown excellent results in advanced colorectal cancer patients who have certain genetic characteristics called 'mismatch repair deficiency (MMR-d)' and 'high microsatellite instability (MSI-h)'. The benefits of immunotherapy as a treatment prior to surgery to remove the tumour (neoadjuvant treatment) has been observed in both melanoma and in glioblastoma with enhanced local and systemic anti-tumour responses.

Pembrolizumab is an immunotherapy drug and works by helping the body's own immune system to fight the cancer cells. The NEOPRISM-CRC trial will investigate whether giving pembrolizumab before surgery is safe, whether it improves the chances of the tumour being removed completely and whether it delays or prevents the cancer from coming back.

Pembrolizumab treatment lasts for a maximum of 9 weeks (maximum of 3 cycles of treatment, each cycle consisting of 3 weeks) and is given prior to surgery. Following surgery patients will be followed up for at least 3 years after their surgery and to a maximum of 5 years. Target recruitment is 78 patients and recruitment is expected to take place over a 42 month period.

Blood, tissue, mouth swabs and stool samples will be collected from patients throughout the trial to better understand the biology of immunotherapy as a treatment for CRC prior to surgery.

DETAILED DESCRIPTION:
The NEOPRISM-CRC study is a phase II clinical trial. The purpose of the trial is to evaluate the efficacy and safety of pembrolizumab (Study IMP) in patients with high risk Stage 2 or Stage 3 MMR-deficient colorectal cancer stratified with tumour mutation burden status.

Pembrolizumab is a type of immunotherapy that has demonstrated excellent results in clinical trials for patients with advanced colorectal cancer who have certain genetic characteristics (mismatch repair deficiency (MMR-d) / high microsatellite instability (MSI-H)). There are previous studies providing evidence that checkpoint inhibitors when given before surgery have shown better local and systemic anti-tumour responses in melanoma and glioblastoma than surgery alone. The main question the researcher wants to investigate is whether pembrolizumab given prior to having surgery delays or prevents the cancer from coming back in advanced colorectal cancer patients with MSI-H or MMR-d. The trial will investigate whether the treatment is safe, whether it improves pathological complete response rate and whether it improves the chances of the tumour being removed completely. The trial will also investigate whether pembrolizumab causes any delay to surgery due to side effects. The trial will also measure post-surgery complications and impact of the treatment on patient's quality of life.

Once patients have enrolled into the NEOPRISM-CRC trial, if patient has consented to a trial colonoscopy, tissue samples will be taken during the procedure and shipped to the FoundationOne Medicine testing Laboratory and analysed to determine the TMB (tumour mutation burden) status assessed by the FOUNDATIONONE®CDx (FM1 Solid CDx) test. If patient does not consent to Trial Colonoscopy, blood sample will be taken to test the TMB status assessed by the FOUNDATIONONE® Liquid CDx (FM1 Liquid CDx) test . In addition if a patient has consented to Trial Colonoscopy, a PCR (Polymerase Chain reaction) test or Microsatellite testing will be done on tissue sample to confirm the Microsatellite Instability (MSI) status.

Patients will receive one of two pre-operative regimens depending upon their TMB status/MSI status

All patients will have one cycle of pembrolizumab 200 mg IV (a cycle is 21 days). Prior to cycle 2 the FM1 result should be available and patients will continue their treatment as follows:

* If results is TMB-high or medium (or MSI-h if FM1 Solid CDx/ Liquid CDx test is not evaluable): A further two cycles of pembrolizumab 200 mg IV every 21 days and then will proceed to surgery 4 - 6 weeks after last dose of pembrolizumab
* If result is TMB-low (or if FM1 Solid CDx/ Liquid CDx test and MSI result are not evaluable): No further cycles of pembrolizumab; will proceed to surgery 4 - 6 weeks after last dose of pembrolizumab

Following surgery, patients will receive standard of care adjuvant treatment which may include post-operative chemotherapy in accordance with investigators clinical decision. Patients will continue to be followed up according to routine standard of care for a maximum of 5 years after surgery.

Target recruitment is 78 patients and recruitment is expected to take place over a 42 month period.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven adenocarcinoma of the colon or rectum which is MMR-d by IHC or MSI-H by PCR (or microsatellite testing if routine practice).
2. Patient is fit (ECOG 0-1) and eligible for planned curative surgery in keeping with NICE guidelines and considered fit/suitable for adjuvant chemotherapy as per local site investigator's discretion based on:

   1. Radiological node positive T1-4 CRC or
   2. Node negative high risk T3 defined as EITHER ≥ 5mm of extramural depth of invasion OR unequivocal EMVI on imaging (regardless of depth) or Node negative T4 disease
3. Patients with rectal cancer are eligible if it is determined that neoadjuvant chemo-radiotherapy is not required to achieve a R0 resection.
4. Patients presenting with acute colonic obstruction may enter the trial only after obstruction is relieved by a successful defunctioning stoma/stent, and when recovered to a fitness level consistent with the other eligibility criteria
5. Adequate bone marrow function:

   * White Blood Cell >3.0 x 10^9/L;
   * Absolute neutrophil count ≥1.5 x 10^9/L
   * Platelets ≥100 x 10^9/L.
   * Haemoglobin ≥90 g/L
6. Adequate renal function:

   GFR >50 mL/min estimated using validated creatinine clearance calculation (e.g. Cockroft-Gault) NB If the calculated creatinine clearance is < 50 mL/min, a formal 24 hour urine collection or isotope clearance must be carried out demonstrating GFR ≥ 50 mL/min as per institutional standards
7. Adequate liver function:

   Total bilirubin < 1.5 times Upper Limit of Normal (ULN) OR direct bilirubin ≤ULN for participants with total bilirubin levels >1.5 × ULN

   AST and ALT ≤ 2.5 × ULN
8. Adequate coagulation:

   International normalized ratio (INR) OR prothrombin time (PT) and Activated partial thromboplastin time (aPTT) ≤1.5 × ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants
9. Aged ≥18 years
10. Able and willing to provide written informed consent
11. Female patients of child bearing potential must be willing to use highly effective contraception for the duration of trial treatment and for 120 days after last dose of pembrolizumab

Exclusion Criteria:

1. Any patient for whom radiotherapy is advised by the MDT
2. Strong evidence of distant metastases or peritoneal nodules (M1)
3. Prior therapy with an anti-PD-1, anti-PD-L1 or anti-PD-L2 agent, or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g. CTLA-4, OX-40, CD137)
4. Prior systemic anti-cancer therapy including investigational agents within 4 weeks prior to registration.

   (NB: Participants must have recovered from all AEs due to previous therapies to ≤Grade 1 or baseline, with the exception of alopecia. Participants with ≤Grade 2 neuropathy may be eligible.) (NB: If participant received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment.)
5. Has received a live vaccine or live-attenuated vaccine within 30 days prior to registration (seasonal flu vaccines that do not contain live virus are permitted). Administration of killed vaccines is allowed
6. Any investigational agents or investigational devices within 4 weeks prior to registration Note: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent.
7. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (dosing exceeding 10mg daily of prednisolone or equivalent), or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment Note: the use of physiologic doses of corticosteroids may be approved after consultation with UCL CTC.
8. Patients with concurrent or previous malignancy that could compromise assessment of the primary or secondary endpoints of the trial
9. Has known active CNS metastases and/or carcinomatous meningitis.
10. Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or to any of its excipients.
11. Has previous severe or life-threatening skin adverse reaction with other immune-stimulatory anticancer agents
12. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs).

    NB: Replacement therapy (e.g. levothyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is permitted.
13. History of (non-infectious) pneumonitis/interstitial lung disease that required steroids, or current pneumonitis/interstitial lung disease
14. Active infection requiring systemic therapy
15. Known history of Human Immunodeficiency Virus (HIV). NB: Testing for HIV for the NEOPRISM-CRC trial is not mandatory, however if this test has been done the result should be known prior to registration.
16. Known active infection for hepatitis B (hepatitis B surface antigen [HbsAg] reactive) or known active hepatitis C (defined as hepatitis C virus [HCV] RNA [qualitative] is detected)

    * Testing is required to determine eligibility. Hepatitis C antibody testing is allowed for initial screening purposes in sites where HCV RNA is not part of standard of care.
    * Patients who are HbsAg positive are eligible if they have received HBV antiviral therapy for at least 4 weeks and have undetectable HBV viral load prior to registration. Participants should remain on anti-viral therapy throughout trial treatment and follow local guidelines for HBV anti-viral therapy post completion of trial treatment.
    * Patients with history of HCV infection are eligible if HCV viral load is undetectable at screening and have completed anti-viral therapy at least 4 weeks prior to registration.
17. Known history of active TB (Mycobacterium tuberculosis).
18. Has had an allogenic tissue/solid organ transplant.
19. Has peritonitis (secondary to perforated tumour)
20. Has a colonic obstruction that has not been defunctioned or stented
21. History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
22. Known psychiatric or substance abuse disorder that would interfere with the participant's ability to cooperate with the requirements of the study.
23. Female patients of child bearing potential who is pregnant or breastfeeding, or expecting to conceive within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of pembrolizumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2022-07-20 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Relapse-free survival | From registration to any signs or symptoms of the cancer or death assessed up to a maximum of 3 years from surgery date
  Relapse-free Survival (RFS) is defined as time from start of treatment to time of any signs or symptoms of the cancer or time of death from any cause.

SECONDARY OUTCOMES:
Pathological complete response rate (pCR) | Pathological complete response rate (pCR) assessed at 3 months following surgery
  A pCR will be defined as having no residual cancer cells in the resected specimen at surgery. Patients who do not achieve pCR or who do not proceed to resectional surgery for any reason will be counted as non-responders.
Overall survival | From registration to death from any cause, assessed up to a maximum of 3 years from surgery date
  Overall survival (OS) is defined as the time from start of treatment to time of death from any cause.
Frequency and severity of adverse events | From informed consent to 3 months after surgery
  Adverse events recorded continuously in relation to each treatment cycle graded using CTCAE criteria
Rate of R0 resection and completed surgery | Assessed from surgery to 28-35 days following surgery
  The incidence of resection types (R0, R1 and R2) will be presented in tables using frequencies, as well as the rate of surgery completed.
Frequency and severity of post-operative surgical complications | Assessed from surgery up to last follow up visit (maximum of 5 years from date of surgery)
  The incidence of surgical complications will be described in tables by complication type/grade using frequencies using the Clavien-Dindo grading system.
Health-related Quality of Life (QoL) and functional outcome | From informed consent to 28-35 days following surgery
  The European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) will be used. The EORTC QLQ-C30 comprises 30 items (i.e. single questions), 24 of which are aggregated into nine multi-item scales, that is, five functioning scales (physical, role, cognitive, emotional and social), three symptom scales (fatigue, pain and nausea/vomiting) and one global health status scale. The remaining six single-item (dyspnoea, appetite loss, sleep disturbance, constipation, diarrhoea and the financial impact) scales assess symptoms. All of the scales and single-item measures range in score from 0 to 100. Higher score for the functioning scales and global health status denote a better level of functioning (i.e. a better state of the patient), while higher scores on the symptom and single-item scales indicate a higher level of symptoms (i.e. a worse state of the patient).
Health-related Quality of Life (QoL) and functional outcome | From informed consent to 28-35 days following surgery
  The EuroQol- 5 Dimension (EQ-5D) will be used. Each dimension in the EQ-5D has five response levels: no problems (Level 1); slight; moderate; severe; and extreme problems (Level 5). Lower score indicates better health, whereas higher score indicate more severe or frequent problems.

CONTACTS AND LOCATIONS:
Overall Officials: Kai-Keen Shiu, Principal Investigator — University College London Hospitals
Locations (5):
- United Kingdom (5):
  - Beatson West of Scotland Cancer Centre, Glasgow
  - St James University Hospital (SJUH), Leeds
  - University College Hospital, London
  - Christie Hospital NHS Trust, Wilmslow Road,, Manchester
  - Southampton General Hospital, Southampton